CLINICAL TRIAL: NCT01468831
Title: A Pilot Study for the Evaluation of Minocycline as a Microglia Inhibitor in the Treatment of Branch Retinal Vein Occlusions
Brief Title: Minocycline to Treat Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110263; 11-EI-0263
Record Dates: First submitted 2011-10-08; First posted 2011-11-10 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-10

CONDITIONS: Retinal Vein Occlusion
Keywords: Minocycline; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; cyclopia sequence; Macular Edema | interventions — Minocycline; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants injected with bevacizumab for three months followed by PRN dosing and placebo twice daily for 24 months
  Interventions: Other: Placebo; Drug: Bevacizumab
- Minocycline (Experimental): Participants injected with bevacizumab for three months followed by PRN dosing and 100mg minocycline twice daily for 24 months
  Interventions: Drug: Minocycline; Drug: Bevacizumab

INTERVENTIONS:
Drug: Minocycline — 100 mg of minocycline in a pink opaque capsule
  Arms: Minocycline
Other: Placebo — Pill with inactive ingredients in a pink opaque capsule
  Arms: Placebo
Drug: Bevacizumab — 1.25 mg bevacizumab injection

SUMMARY:
Background:

- Branch retinal vein occlusion (BRVO) is a blockage of the small veins that carry blood away from the retina in the back of the eye. It often leads to macular edema, a swelling of the retina that is a common source of vision loss. Studies suggest that inflammation might be a cause. Minocycline is a drug that might help prevent cells involved in inflammation from becoming activated. It is approved for use as an antibiotic, but it has not yet been tested to see if it can treat BRVO.

Objectives:

- To test the safety and effectiveness of minocycline as a treatment for branch retinal vein occlusion.

Eligibility:

- Individuals at least 18 years of age who have branch retinal vein occlusion in at least one eye, with vision between 20/32 and 20/200.

Design:

* This study lasts 2 years, with at least 25 visits.
* Participants will be screened with a physical exam and medical history. They will also have blood tests and an eye exam. One eye will be selected as the study eye to receive the medicine.
* Those in the study will take minocycline or a placebo pill twice a day, about 12 hours apart, for 2 years.
* Participants will have monthly visits for blood tests and full eye exams to study the effect of the treatment. Other exams may include thyroid tests and eye imaging studies. Those in the study may also receive injections of a drug to prevent the growth of new blood vessels in the eye.

DETAILED DESCRIPTION:
Objective:

Retinal vein occlusions (RVO) are significant sources of vision loss, affecting mostly healthy people over 55 years of age. The common source of vision loss is the macular edema accompanying the retinal injury. Very recently, studies employing monthly anti-vascular endothelial growth factor (VEGF) treatments have demonstrated a benefit to this line of treatment; however, the duration of effectiveness appears to be short lived and the length of time needed for these monthly injections remains unknown. A histologic study of human retinas with RVOs found the presence of activated microglia. Microglia are capable of migrating through the retina to sites of inflammation to associate closely with neurons and the vasculature, and are key cellular players in the mediation of processes of chronic inflammation. For these reasons, microglia represent a promising cellular target for forms of therapy that limit the deleterious inflammatory changes found in vein occlusions. Minocycline, a second-generation tetracycline, has been shown to exhibit anti-inflammatory properties, including microglia inhibition. The objective of this study is to investigate the safety and efficacy of minocycline as a microglia inhibitor in participants with branch retinal vein occlusion (BRVO).

Study Population:

A minimum of ten and a maximum of 20 participants who meet the eligibility criteria may be enrolled. Eligibility criteria include: foveal center-involved macular edema secondary to a BRVO, retinal thickness in the central subfield greater than 350 microns as measured by optical coherence tomography (OCT) and visual acuity (VA) between 20/32 and 20/200 in the study eye.

Design:

In this pilot, double-masked, randomized, multi- center study, participants will receive monthly bevacizumab injections for the first three months, followed by PRN dosing. In addition, participants will take an oral dose of 100 mg of minocycline or placebo twice daily for 24 months. During each monthly visit, participants will have their visual acuity measured and will undergo OCT testing to measure retinal thickness. At the Month 3 visit and thereafter, participants will be evaluated for "improvement" and "worsening" and will be eligible for additional bevacizumab treatment and/or investigational product (IP) depending on which criteria they fulfill. Additionally, at Month 12, participants will also be evaluated for no improvement.

Outcome Measures:

The primary outcome is the difference in mean change in best-corrected visual acuity (BCVA), as measured in ETDRS letters, between the minocycline and placebo groups in the study eye at 12 months compared to baseline. Secondary outcomes include the difference between the minocycline and placebo groups in the number of intravitreal bevacizumab injections between 12 and 24 months and baseline, changes in mean macular sensitivity as measured by microperimetry at 3, 6, 12, 18 and 24 months compared to baseline, the mean change in BCVA at 24 months compared to baseline, the changes in retinal thickness as measured by OCT at 6, 12, 18 and 24 months compared to baseline, number of participants improving greater than or equal to 1 logOCT scale step at 12 and 24 months compared to baseline, as well as changes in fluid leakage in the macula as demonstrated by fluorescein angiography at 12 and 24 months compared to baseline. Safety outcomes include the number of participant withdrawals, the number and severity of systemic and ocular toxicities and the number of adverse events.

ELIGIBILITY:
PARTICIPANT ELIGIBILITY CRITERIA

INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable:

1. Participant is 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Female participants of childbearing potential must not be pregnant or breast-feeding and must be willing to undergo serum (BRC sites only) and urine pregnancy tests throughout the study.
4. Female participants of childbearing potential and male participants able to father children must meet the following site-specific criteria:

   1. For the NEI Site: Female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for one week after study medication discontinuation (based on the half life of minocycline which is 11-22 hours). Acceptable methods of contraception include:

      * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
      * intrauterine device,
      * barrier methods (diaphragm, condom) with spermicide, or
      * surgical sterilization (hysterectomy or tubal ligation).
      * Note: Oral birth control pills must be used with caution as minocycline decreases the effectiveness of some oral contraceptives. Participants already taking oral contraceptives may continue to use them, but must agree to use at least one other method of birth control while on study.
   2. For the BRC Sites: Female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, or be completely abstinent from intercourse. Male participants or male partners (of female participants) who have not had a vasectomy or are not abstinent are required to use a condom with spermicide throughout the course of the study and for one week after study medication discontinuation (based on the half life of minocycline which is 11-22 hours). Female participants of childbearing potential or female partners (of male participants) of childbearing potential must practice one of the below acceptable methods of contraception throughout the course of the study and for one week after study medication discontinuation:

      * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
      * intrauterine device,
      * barrier methods (e.g., diaphragm) with spermicide, or
      * surgical sterilization (hysterectomy or tubal ligation).
      * Notes: i) Abstinence is only acceptable when it is the participant's preferred and usual lifestyle choice. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. ii) Oral birth control pills must be used with caution as minocycline decreases the effectiveness of some oral contraceptives. Participants already taking oral contraceptives may continue to use them, but must agree to use at least one other method of birth control while on study. iii)) It should be noted that two forms of contraception (as specified above) will be used by sexually active participants for the duration of the study and for one week after study medication discontinuation.
5. Participants must agree to notify the study investigator or coordinator if any of their doctors initiate a new medication during the course of the study.
6. Participant must have normal renal function and liver function or have mild abnormalities not above grade 1 as defined by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
7. Participant must agree to minimize exposure to sunlight or artificial UV rays and to wear protective clothing, sunglasses and sunscreen (minimum SPF 15) if s/he must be out in the sun.
8. Participant has at least one eye that meets the study eye criteria.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present:

1. Participant is in another investigational study and actively receiving investigational product for BRVO.
2. Participant is unable to comply with study procedures or follow-up visits.
3. Participant has a known hypersensitivity to sodium fluorescein dye.
4. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
5. Participant has a history of chronic renal failure requiring dialysis or kidney transplant.
6. Participant has a history of chronic hepatitis or liver failure.
7. Participant has an allergy or hypersensitivity to minocycline or any drug in the tetracycline family.
8. Participant is currently taking a tetracycline medication.
9. Participant is taking any medication that could adversely interact with minocycline such as methoxyflurane.
10. Participant has a blood pressure of greater than 180/110 (systolic above 180 OR diastolic above 110).

    a. If blood pressure is brought below 180/110 by anti-hypertensive treatment, the participant can become eligible.
11. Participant is currently being treated with systemic anti-VEGF agents or systemic steroids.
12. Participant had a cerebral vascular event (CVA) or myocardial infarction (MI) within three months prior to study entry.
13. Participant has a history of thyroid cancer.

STUDY EYE ELIGIBILITY CRITERIA:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below:

STUDY EYE INCLUSION CRITERIA

1. The study eye has a best-corrected ETDRS visual acuity score between 78 and 34 letters (i.e., between 20/32 and 20/200).
2. The study eye shows evidence of definite retinal thickening due to a BRVO based on clinical examination involving the center of the macula that is not refractory to further therapy as based on the investigator's clinical judgment. BRVO is defined as an eye that had retinal hemorrhage or other biomicroscopic evidence of RVO (e.g., telangiectatic capillary bed) and a dilated (or previously dilated) venous system in one or two quadrants or less of the retina drained by the affected vein. Hemiretinal vein occlusion (HRVO) is an RVO that involves two altitudinal quadrants. In this study, eyes with a HRVO will be considered a BRVO and are given the same treatment as BRVO eyes.
3. The study eye has retinal thickness in the central subfield on baseline OCT measurement >350 microns, as measured by Zeiss Cirrus spectral domain OCT, or an equivalent retinal thickness on a similar OCT machine.
4. The study eye has media clarity and pupillary dilation sufficient for adequate fundus photographs. Furthermore, the participant must be able to cooperate during the procedure for accurate fundus photographs.

STUDY EYE EXCLUSION CRITERIA

1. The study eye has macular edema considered to be due to a cause other than BRVO.
2. An eye should not be considered eligible if:

   1. The macular edema is considered to be related to cataract extraction, or
   2. Clinical examination and/or OCT suggest that vitreoretinal interface disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of the macular edema, or
   3. Clinical examination, medical history and/or fluorescein angiography suggest that diabetic retinopathy is the primary cause of the edema.
   4. The study eye has a history of a recurrent RVO.
   5. The study eye has a history of RVO present for > 18 months.
   6. A brisk afferent pupillary defect (APD) is present in the study eye.
   7. An ocular condition is present in the study eye such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, laser scar at fovea, non-retinal condition).
   8. An ocular condition (other than RVO) is present that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
   9. A substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal) is present in the study eye.
   10. The study eye has had panretinal or sectoral scatter photocoagulation (PRP) within four months prior to study entry.
   11. The study eye has had pars plana vitrectomy within six months prior to study entry.
   12. The study eye has undergone major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within three months prior to study entry.
   13. A yttrium aluminum garnet (YAG) capsulotomy has been performed on the study eye within two months prior to study entry.
   14. The study eye has had treatment < 3 months prior to study entry of intravitreal or periocular steroid injections.
   15. The study eye has had treatment < 28 days prior to study entry of intravitreal anti-VEGF agents.

STUDY EYE SELECTION CRITERIA IN CASES OF BILATERAL DISEASE

If both eyes of a participant meet the criteria, the study eye will be determined at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Cukras, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Bristol Eye Hospital, Bristol, United Kingdom

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-EI-0263.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recriutment was activated on November 18, 2011 at the NEI site and on May 25, 2018 at the BEH site. Enrollment was closed on May 13, 2019 at the NEI site and on December 31, 2019 at the BEH site.
Units Other Than Participants: Eye
Period: Overall Study
Arm/Group | Placebo | Minocycline
Started | 4; 4 Eye | 5; 5 Eye
Month 12 (Primary Outcome) | 4; 4 Eye | 4; 4 Eye
Completed | 4; 4 Eye | 4; 4 Eye
Not Completed | 0; 0 Eye | 1; 1 Eye

BASELINE CHARACTERISTICS:
Population: Study eye is the unit of analysis and is chosen based on study eye inclusion/exclusion criteria. If both eyes of a participant meet the criteria, the study eye will be determined at the investigator's discretion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Minocycline | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.21) | 70.6 (5.55) | 67.0 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7
  United Kingdom | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best-corrected Visual Acuity (BCVA) in the Study Eye at 12 Months Compared to Baseline.
Description: The primary outcome measure is the mean difference between the minocycline and placebo groups in the change in best-corrected visual acuity (BCVA), as measured in ETDRS letters, in the study eye at 12 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 12 months.
Time Frame: Baseline to Month 12
Population: The primary outcome analysis population includes those participants who were exposed to IP and were followed up for at least 12 months. One participant in the minocycline group was excluded from the analysis because their Month 12 data was not recorded due to their withdrawal from the study prior to Month 12.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
ETDRS letters | 5.3 (9.6) | 13.0 (11.3)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo arms in change in BCVA in the study eye at Month 12 compared to baseline is reported; Mean Difference (Net) = 7.8, 95% CI 2-sided [-10.6 to 26.1], Standard Deviation 7.4 — Difference = Minocycline - Placebo

2. Secondary Outcome: Number of Bevacizumab Injections From Baseline to 12 Months
Description: The outcome measure is the difference between the minocycline and placebo groups in the number of bevacizumab injections administered to participants between baseline and 12 months.
Time Frame: Baseline to Month 12
Population: The secondary outcomes are based on the safety population, which includes all participants who were exposed to IP, regardless of adherence to protocol.
Measure: Mean (Standard Deviation); unit: bevacizumab injections
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 5
bevacizumab injections | 5.5 (1.9) | 6.6 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo treatment arms in number of bevacizumab injections received from baseline to Month 12 is reported; Mean Difference (Net) = 1.1, Standard Deviation 1.4 — Difference = Minocycline - Placebo

3. Secondary Outcome: Number of Bevacizumab Injections From Baseline to 24 Months
Description: The outcome measure is the difference between the minocycline and placebo groups in the number of bevacizumab injections administered to participants between baseline and 24 months.
Time Frame: Baseline to Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bevacizumab injections
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 5
bevacizumab injections | 9.0 (5.9) | 8.8 (4.2)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; The mean difference between the minocycline and placebo treatment arms in number of bevacizumab injections received from baseline to Month 24 is reported; Test type: Other; Mean Difference (Net) = -0.2, Standard Deviation 3.5 — Difference = Minocycline - Placebo

4. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye as Measured by Microperimetry at 3 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in macular sensitivity as measured by microperimetry in the study eye at 3 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 3 months. Higher macular sensitivity (higher db) is better.
Time Frame: Baseline to Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: db
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 5
db | 0.5 (1.2) | -0.4 (2.5)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo groups in the change in macular sensitivity in the study eye at Month 3 compared to baseline is reported; Mean Difference (Net) = -0.8, 95% CI 2-sided [-3.9 to 2.3], Standard Deviation 1.3 — Difference = Minocycline - Placebo

5. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye as Measured by Microperimetry at 6 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in macular sensitivity as measured by microperimetry in the study eye at 6 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 6 months. Higher macular sensitivity (higher db) is better.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: db
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 5
db | 0.7 (1.3) | -1.5 (1.7)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo groups in the change in macular sensitivity in the study eye at Month 6 compared to baseline is reported; Mean Difference (Net) = -2.1, 95% CI 2-sided [-4.5 to 0.3], Standard Deviation 1.0 — Difference = Minocycline - Placebo

6. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye as Measured by Microperimetry at 12 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in macular sensitivity as measured by microperimetry in the study eye at 12 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 12 months. Higher macular sensitivity (higher db) is better.
Time Frame: Baseline to Month 12
Population: The secondary outcomes are based on the safety population, which includes all participants who were exposed to IP, regardless of adherence to protocol. One participant in the minocycline group was excluded because their Month 12 data was not recorded due to withdrawal from the study prior to the Month 12 visit.
Measure: Mean (Standard Deviation); unit: db
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
db | 1.1 (1.4) | -1.4 (3.3)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo groups in the change in macular sensitivity in the study eye at Month 12 compared to baseline is reported; Mean Difference (Net) = -2.5, 95% CI 2-sided [-7.5 to 2.5], Standard Deviation 1.8 — Difference = Minocycline - Placebo

7. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye as Measured by Microperimetry at 18 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in macular sensitivity as measured by microperimetry in the study eye at 18 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 18 months. Higher macular sensitivity (higher db) is better.
Time Frame: Baseline to Month 18
Population: The secondary outcomes are based on the safety population, which includes all participants who were exposed to IP, regardless of adherence to protocol. Two participants in the minocycline group was excluded due to missing macular sensitivity data at Month 18.
Measure: Mean (Standard Deviation); unit: db
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 3
db | 0.4 (3.0) | -3.1 (2.9)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo groups in the change in macular sensitivity in the study eye at Month 18 compared to baseline is reported; Mean Difference (Net) = -3.5, 95% CI 2-sided [-9.4 to 2.4], Standard Deviation 2.2 — Difference = Minocycline - Placebo

8. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye as Measured by Microperimetry at 24 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in macular sensitivity as measured by microperimetry in the study eye at 24 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 24 months. Higher macular sensitivity (higher db) is better.
Time Frame: Baseline to Month 24
Population: The secondary outcomes are based on the safety population, which includes all participants who were exposed to IP, regardless of adherence to protocol. One participant in the minocycline group was excluded because their Month 24 data was not recorded due to withdrawal from the study prior to the Month 24 visit.
Measure: Mean (Standard Deviation); unit: db
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
db | 0.1 (3.2) | -3.7 (3.5)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo groups in the change in macular sensitivity in the study eye at Month 24 compared to baseline is reported; Mean Difference (Net) = -3.7, 95% CI 2-sided [-9.5 to 2], Standard Deviation 2.4 — Difference = Minocycline - Placebo

9. Secondary Outcome: Mean Change in the ETDRS BCVA in the Study Eye at 24 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in best-corrected visual acuity (BCVA), as measured in ETDRS letters, in the study eye at 24 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 24 months.
Time Frame: Baseline to Month 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
ETDRS letters | 2.8 (10.7) | 8.5 (14.8)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo arms in change in BCVA in the study eye at Month 24 compared to baseline is reported; Mean Difference (Net) = 5.8, 95% CI 2-sided [-17.1 to 28.6], Standard Deviation 9.1 — Difference = Minocycline - Placebo

10. Secondary Outcome: Changes in Retinal Thickness in the Study Eye as Measured by Optical Coherence Tomography (OCT) at 6 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in central retinal thickness in the study eye at 6 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 6 months.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 5
micrometers | -91.0 (53.8) | -142.8 (146.5)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo treatment arms in change in retinal thickness as measured by OCT in the study eye at Month 6 compared to baseline is reported; Mean Difference (Net) = -51.8, 95% CI 2-sided [-231.2 to 127.6], Standard Deviation 70.8 — Difference = Minocycline - Placebo

11. Secondary Outcome: Changes in Retinal Thickness in the Study Eye as Measured by Optical Coherence Tomography (OCT) at 12 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in central retinal thickness in the study eye at 12 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 12 months.
Time Frame: Baseline to Month 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
micrometers | -99.3 (45.0) | -144.8 (303.7)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo treatment arms in change in retinal thickness as measured by OCT in the study eye at Month 12 compared to baseline is reported; Mean Difference (Net) = -45.5, 95% CI 2-sided [-522.6 to 431.6], Standard Deviation 153.5 — Difference = Minocycline - Placebo

12. Secondary Outcome: Changes in Retinal Thickness in the Study Eye as Measured by Optical Coherence Tomography (OCT) at 18 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in central retinal thickness in the study eye at 18 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 18 months.
Time Frame: Baseline to Month 18
Population: The secondary outcomes are based on the safety population, which includes all participants who were exposed to IP, regardless of adherence to protocol. One participant in the minocycline group was excluded because their Month 18 data was not recorded due to withdrawal from the study prior to the Month 18 visit.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
micrometers | -111.8 (63.9) | -124.5 (321.3)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo treatment arms in change in retinal thickness as measured by OCT in the study eye at Month 18 compared to baseline is reported; Mean Difference (Net) = -12.8, 95% CI 2-sided [-513.1 to 487.6], Standard Deviation 163.8 — Difference = Minocycline - Placebo

13. Secondary Outcome: Changes in Retinal Thickness in the Study Eye as Measured by Optical Coherence Tomography (OCT) at 24 Months Compared to Baseline
Description: The outcome measure is the mean difference between the minocycline and placebo groups in the change in central retinal thickness in the study eye at 24 months compared to baseline. Values presented represent mean and standard deviation of change from baseline at 24 months.
Time Frame: Baseline to Month 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
micrometers | -125.8 (63.4) | -135.3 (307.0)
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The mean difference between the minocycline and placebo treatment arms in change in retinal thickness as measured by OCT in the study eye at Month 24 compared to baseline is reported; Mean Difference (Net) = -9.5, 95% CI 2-sided [-487 to 468], Standard Deviation 156.8 — Difference = Minocycline - Placebo

14. Secondary Outcome: Number of Participants Improving ≥ 1 logOCT Scale Step in the Study Eye at 12 Months Compared to Baseline
Description: The outcome measure is the difference between the minocycline and placebo groups in the number of participants experiencing an improvement of ≥ 1 logOCT scale step from baseline to Month 12. Improvement in ≥ 1 logOCT scale step is defined as a decrease of ≥ 1-step on the logOCT scale. A 1-step decrease is equivalent to at least a 20% improvement of central macular thickness.
Time Frame: Baseline to Month 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
Participants | 2 | 3
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The difference between the minocycline and placebo treatment arms in number of participants improving ≥ 1 logOCT scale step in the study eye at Month 12 compared to baseline is reported; Difference in Number of Participants = 1 — Difference = Minocycline - Placebo

15. Secondary Outcome: Number of Participants Improving ≥ 1 logOCT Scale Step in the Study Eye at 24 Months Compared to Baseline
Description: The outcome measure is the difference between the minocycline and placebo groups in the number of participants experiencing an improvement of ≥ 1 logOCT scale step from baseline to Month 24. Improvement in ≥ 1 logOCT scale step is defined as a decrease of ≥ 1-step on the logOCT scale. A 1-step decrease is equivalent to at least a 20% improvement of central macular thickness.
Time Frame: Baseline to Month 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
Participants | 3 | 3
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The difference between the minocycline and placebo treatment arms in number of participants improving ≥ 1 logOCT scale step in the study eye at Month 24 compared to baseline is reported; Difference in Number of Participants = 0 — Difference = Minocycline - Placebo

16. Secondary Outcome: Number of Participants Experiencing Changes in Fluid Leakage in the Macula of the Study Eye as Demonstrated by Fluorescein Angiography at 12 Months Compared to Baseline
Description: The outcome measure is the difference between the between the minocycline and placebo groups in the number of participants experiencing changes in fluid leakage in the macula of the study eye as demonstrated by fluorescein angiography at 12 months compared to baseline. The counts presented are the number of participants experiencing decrease, increase, or no change in fluid leakage from baseline.
Time Frame: Baseline to Month 12
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
participants
  Decrease | 4 | 2
  Increase | 0 | 0
  No Change | 0 | 2
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The difference between the minocycline and treatment arms in the number of participants experiencing a decrease in fluid leakage at Month 12 compared to baseline is reported; Difference in Number of Participants = -2 — Difference = Minocycline - Placebo
Statistical Analysis 2: Comparison: Placebo vs Minocycline; Test type: Other — The difference between the minocycline and treatment arms in the number of participants experiencing an increase in fluid leakage at Month 12 compared to baseline is reported; Difference in Number of Participants = 0 — Difference = Minocycline - Placebo
Statistical Analysis 3: Comparison: Placebo vs Minocycline; Test type: Other — The difference between the minocycline and treatment arms in the number of participants experiencing no change in fluid leakage at Month 12 compared to baseline is reported; Difference in Number of Participants = 2 — Difference = Minocycline - Placebo

17. Secondary Outcome: Number of Participants Experiencing Changes in Fluid Leakage in the Macula of the Study Eye as Demonstrated by Fluorescein Angiography at 24 Months Compared to Baseline.
Description: The outcome measure is the difference between the between the minocycline and placebo groups in the number of participants experiencing changes in fluid leakage in the macula of the study eye as demonstrated by fluorescein angiography at 24 months compared to baseline. The counts presented are the number of participants experiencing decrease, increase, or no change in fluid leakage from baseline.
Time Frame: Baseline to Month 24
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo | Minocycline
Number analyzed (Participants) | 4 | 4
participants
  Decrease | 4 | 3
  Increase | 0 | 1
  No Change | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Minocycline; Test type: Other — The difference between the minocycline and treatment arms in the number of participants experiencing a decrease in fluid leakage at Month 24 compared to baseline is reported; Difference in Number of Participants = -1 — Difference = Minocycline - Placebo
Statistical Analysis 2: Comparison: Placebo vs Minocycline; Test type: Other — The difference between the minocycline and treatment arms in the number of participants experiencing an increase in fluid leakage at Month 24 compared to baseline is reported; Difference in Number of Participants = 1 — Difference = Minocycline - Placebo
Statistical Analysis 3: Comparison: Placebo vs Minocycline; Test type: Other — The difference between the minocycline and treatment arms in the number of participants experiencing no change in fluid leakage at Month 24 compared to baseline is reported; Difference in Number of Participants = 0 — Difference = Minocycline - Placebo

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Placebo | Minocycline
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Minocycline (N=5)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) — CRVO OS
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Minocycline (N=5)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral mucosal discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (4) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
Renal function test abnormal (Investigations) | 1 (1) | 0 (0)
Thyroid function test abnormal (Investigations) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 1 (1)
Retinal pigmentation (Eye disorders) | 0 (0) | 1 (1) — Natural progression of disease
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (2) — Natural progression of disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT01468831/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT01468831/SAP_001.pdf
  • Informed Consent Form (2019-02-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT01468831/ICF_002.pdf